CLINICAL TRIAL: NCT04458376
Title: Internet-based Self-help Program for Vestibular Rehabilitation in Chronic Dizziness; a Pilot Study
Brief Title: Internet-based Self-help Program for Vestibular Rehabilitation in Chronic Dizziness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Møre og Romsdal HF (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 137107
Record Dates: First submitted 2020-06-29; First posted 2020-07-07 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Vertigo
Keywords: Rehabilitation; Telerehabilitation; Internet; Norway
MeSH Terms: conditions — Vertigo

STUDY DESIGN:
Intervention Model Description: Consecutively recruited at Department of Neurology at Molde County hospital, outpatient clinic.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Follows the internet-based self-help program (Experimental)
  Interventions: Behavioral: Internet-based self-help program

INTERVENTIONS:
Behavioral: Internet-based self-help program — The program is divided into six short weekly lessons providing information about chronic dizziness and vestibular rehabilitation, and demonstrating the exercises by video. The program is freely available in the Norwegian electronic handbook for physicians (NEL). The participants in the study will receive the internet address after inclusion in the study.

SUMMARY:
Chronic dizziness,or persistent positional perceptual dizziness (PPPS) is a common condition that results in impaired quality of life and work ability of those affected. Vestibular Rehabilitation (VR) is an evidence-based and recommended treatment for chronic dizziness. The treatment involves training in specific exercises that challenge the balance system and eventually improve dizziness. The main challenge with this treatment is that it is usually best provided with individual follow-up of therapists trained in the method. Limited resources and the lack of dissemination of this knowledge mean that only a minority of patients receive adequate treatment. An internet-based self-help program in vestibular rehabilitation has been developed in Norwegian with demonstration and instructions of exercises. The program has six lessons, together lasting for six weeks. Patients are given the opportunity to exercise at home, without the use of treatment resources and without spending time traveling to the treatment site. Patients will have access through their general practitioner or health institution at no extra cost. If it turns out that the program works according to the intention, the investigators will be able to offer VR to a large number of PPPS patients who previously would not receive treatment for their condition.

The aim of the pilot study is to find out if the internet program for PPPS works as intended and evaluate incoming data and make changes to the program. In addition, the investigators will gain experience in using the program before designing a randomized clinical trial (RCT). The aim of such an RCT would be to compare this internet based treatment to traditional treatment.

ELIGIBILITY:
Inclusion Criteria:

* Satisfy diagnostic criteria for persistent positional perceptual dizziness (PPPS) or satisfy criteria with a duration of <3 months
* Vertigo symptom scale (VSS-SF) >12

Exclusion Criteria:

* Cognitive dysfunction that is so pronounced that it will make participation difficult
* Unable to read, understand Norwegian
* Severe medical or psychiatric illness (including substance abuse) that reduces the patient's ability to follow the VR program

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-02-09 (Actual); Study Completion 2021-02-09 (Actual)

PRIMARY OUTCOMES:
user experience ease of use | 3 months
  semi-structured conversation interview with score tools. The ease of use of the course will be scored in a 7 question questionnaire, rated 1-7 from very good to very bad. The questions are whether the program worked well, was boring, if it was the right dose of exercises, if the text was understandable, instructive, how was the yield and degree of subjective improvement. Participants will also be asked for preparation suggestions.
Symptom change | 3 months
  The Niigata persistent positional perceptual dizziness (PPPD) Questionnaire (NPQ) contains 12 questions in which patients answer questions about provocation from three aggravating factors of PPPD (upright posture / gait, movement and visual stimulation). Each factor is evaluated using questions that score the severity from 0 (none) to 6 (unbearable) ailments
Symptom change | 3 months
  VSS - vertigo symptom score form. Consists of 15 questions. Each answer is scored on a 5-point scale (0-4), and a measure of the severity of the symptoms is obtained by summing. The total score ranges from 0-60, higher scores indicate more serious problems. Severe dizziness is defined as ≥ 12 points on the total scale. The scale includes two subscales: 8 selected questions related to vertigo and balance (score ranging from 0-32), and 7 selected questions related to autonomic anxiety symptoms (score ranging from 0-28)

CONTACTS AND LOCATIONS:
Overall Officials: Torstein Hole, md phd, Study Director — Møre og Romsdal Hospital Trust
Locations (1):
- Molde sykehus, Molde, Norway